CLINICAL TRIAL: NCT03747289
Title: Comparison of the Effect of a Weight Bearing Protocol and a Non-weight Bearing Protocol on Osteoporotic Women With Chronic Low Back Pain
Brief Title: Comparison of a Weight Bearing and a Non-weight Bearing Protocol on Osteoporotic Women With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bait Balev Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0043-18-BBL
Record Dates: First submitted 2018-08-01; First posted 2018-11-20 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-01

CONDITIONS: Osteoporosis; Low Back Pain
MeSH Terms: conditions — Osteoporosis; Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Masking Description: the investigator will check all the participants without knowing to which group they are assigned to
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- weight bearing group (Experimental): performing exercises in a weight bearing posture
  Interventions: Other: performing exercises in a weight bearing posture
- non-weight bearing group (Active Comparator): performing exercises in a non- weight bearing posture
  Interventions: Other: performing exercises in a non weight bearing posture

INTERVENTIONS:
Other: performing exercises in a weight bearing posture — 20 participants will perform exercises in a weight bearing posture
  Arms: weight bearing group
Other: performing exercises in a non weight bearing posture — 20 participants will perform exercises in a non weight bearing posture
  Arms: non-weight bearing group

SUMMARY:
The effect of exercising in different body positions on bone growth in osteoporotic women is known, but its effect on their function, low back pain, lumbar range of motion and quality of life remains unknown. Therefore, the investigators plan to make a comparison of the effect of a weight bearing protocol and a non-weight bearing protocol on osteoporotic women with chronic low back pain.

40 women with osteoporosis and low back pain will be divided into two groups. Each group will be given a specific exercise protocol, twice a week for four weeks, 45 minutes each time. The participants will be tested before starting the program, immediately after finishing it and again two months later. The tests will include filling out the Roland Morris Disability Questionnaire, the SF-36 quality of life Questionnaire, pain measurement by VAS (Visual Analogue Scale) and lumbar range of motion measurement by a digital Inclinometer.

Statistical analysis will be made in order to compare the dependent variables between groups.

DETAILED DESCRIPTION:
40 women with osteoporosis and low back pain will be recruited by referral of doctors to the physical therapy clinic in Bat-Yam, Israel. Each woman will be tested by one investigator after meeting the criteria of eligibility and after obtaining formed consent . The tests will include filling out the Roland Morris Disability Questionnaire, the SF-36 quality of life Questionnaire, pain measurement by VAS and lumbar range of motion measurement by a digital Inclinometer. By order of appearance, each participant will be assigned to one of two groups - weight bearing group or non-weight bearing group. After recruiting at least 3 participants in each group, a different investigator will begin a specific exercise protocol for each of the groups for four weeks - twice a week, 45 minutes each time, a total of 8 sessions. After each participant finishes all 8 sessions, she will be tested for the second time by the first investigator, the same tests as the first time. A third identical test will be preformed two months after finishing the program.

After all the participants finish the program statistical analysis will be made in order to compare the dependent variables between groups.

ELIGIBILITY:
Inclusion Criteria:

* women with osteoporosis (T score lower than -2.5)
* women whom had suffered from non specific low back pain for the last 3 months or more.

Exclusion Criteria:

* history of operations in the spine
* history of cancer or neurologic disease
* history of fractures
* previous trauma to the spine
* persons whom for any reason cannot sit on a chair or lie on a mattress for 45 minutes

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 53 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
Change of physical disability | 3 months
  the Roland Morris Disability Questionnaire. The score of the questionnaire is the total number of items checked - i.e. from a minimum of 0 to a maximum of 24.

SECONDARY OUTCOMES:
change in lumbar range of motion - flexion and extension | 3 months
  digital inclinometer. The change will be assessed by the difference in number of degrees measured
change in pain intensity | 3 months
  Visual Analogue Scale (VAS). A scale from 0 (no pain) to 10 (the worst possible pain)
change in health related quality of life | 3 months
  the Short Form-36 (SF-36) quality of life Questionnaire. A questionnaire of 36 questions, each response receives a specific value

CONTACTS AND LOCATIONS:
Locations (1):
- Maccabi health services, Bat Yam, Israel